CLINICAL TRIAL: NCT01390883
Title: Special Drug Use Investigation for ARIXTRA (Fondaparinux) Abdominal (Urology,Obstetrics,Gynecology)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112721
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fondaparinux

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients prescribed fondaparinux: Patients undergoing abdominal surgery in urology, obstetrics and gynecology departments prescribed fondaparinux during study period
  Interventions: Drug: Fondaparinux Sodium

INTERVENTIONS:
Drug: Fondaparinux Sodium

SUMMARY:
The purpose of this study is to collect and assess information on safety and efficacy of fondaparinux in patients undergoing abdominal surgery in urology, obstetrics and gynecology departments who are at high risk of venous thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing abdominal surgery in urology, obstetrics and gynecology departments

Exclusion Criteria:

* Patients with a history of hypersensitivity to the ingredients of fondaparinux
* Patients with bleeding (bleeding in important organs, sucn as retroperitoneal bleed)
* Patients with acute bacterial endocarditis
* Patients with severe renal impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients undergoing abdominal surgery in urology, obstetrics and gynecology departments who are at high risk of venous thromboembolism
Sampling Method: Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2008-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The number of adverse events in Japanese patients treated with fondaparinux | 4 months at maximum
Presence or absence of venous thromboembolism after treatment of fondaparinux | 4 months at maximum

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline